CLINICAL TRIAL: NCT02736695
Title: Assessment of Hyperphosphorylated Tau PET Binding in Primary Progressive Aphasia and FTD
Brief Title: Assessment of Hyperphosphorylated Tau PET Binding in Primary Progressive Aphasia and Frontotemporal Dementia
Acronym: SLD3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Keith A. Josephs, Professor of Neurology, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-001703; 1R21NS094684-01 (NIH)
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Primary Progressive Aphasia; Behavioral Variant of Frontotemporal Dementia; Frontotemporal Dementia, Behavioral Variant
Keywords: PPA; bvFTD; FTD
MeSH Terms: conditions — Aphasia, Primary Progressive; Pick Disease of the Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tau PET Scan, F-18 AV 1451 (Experimental): All subjects will receive a Tau PET scan.
  Interventions: Drug: F-18 AV 1451
- Normal Controls (No Intervention): Subjects from our NIH funded Mayo Clinic Study of Aging (U01 AG006786) who have completed the identical tau-PET protocol with AV-1451 and MRI and clinical protocols. These participants were not consented or enrolled in this study.

INTERVENTIONS:
Drug: F-18 AV 1451 — Tau binding agent
  Arms: Tau PET Scan, F-18 AV 1451

SUMMARY:
This study is designed to learn more about overall tau burden in the brain of patients with Primary Progressive Aphasia (PPA) and Frontotemporal Dementia.

DETAILED DESCRIPTION:
Primary progressive aphasia (PPA) is an umbrella term that encompasses a group of neurodegenerative syndromes characterized by varying combinations of progressive speech and language problems. Three clinical variants of PPA have been described and are well recognized: the agrammatic variant characterized by grammatical errors in speech and writing and typically associated with phonetic errors in speech; the semantic variant characterized by poor naming from loss of knowledge about the meaning of words; and the logopenic variant characterized by word retrieval problems and poor sentence repetition from impairment of working memory and phonemic errors. Pathological studies of PPA patients that died with postmortem examination of their brains have demonstrated that PPA is associated with a number of different abnormal cellular proteins that do not have perfect associations with the three PPA variants. One such protein is the microtubule associated protein, tau, which is the most common abnormal protein found in the brains of patients with PPA. Tau is an important protein that has been linked to the neurodegenerative process in many diseases. No neuroimaging studies have investigated tau deposition in PPA and hence the binding characteristics of AV-1451 (the Tau binding drug used in this study) in PPA are unknown. Understanding the binding characteristics of AV-1451 is crucial to help determine whether it can serve as a biomarker for tau deposition in the brains of patients with PPA.

FTD or Frontotemporal Dementias, including bvFTD, will also be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Must be over the age of 18
* Must speak English as your primary language
* Must have an informant who can provide independent evaluation of functioning
* Must present with a chief complaint of progressive impairment of speech/language or changes in behavior
* Must fulfill diagnostic criteria for Primary Progressive Aphasia or Frontotemporal Dementia

Exclusion Criteria:

* Any subject who is mute or whose speech is unintelligible will be excluded
* All subjects with concurrent illnesses that could account for speech and language deficits, such as traumatic brain injury, strokes or developmental syndromes, and subjects meeting criteria for another neurodegenerative disease, such as amnestic Alzheimer's type dementia, dementia with Lewy bodies, progressive supranuclear palsy, and corticobasal syndrome will be excluded
* All pregnant, post-partum and breast-feeding women will be excluded
* Subjects will also be excluded if MRI is contraindicated (metal in head, cardiac pace maker, etc.), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma or intracranial neoplasm), or if they are medically unstable or are on medications that might affect brain structure or metabolism,(e.g. chemotherapy).
* Subjects who meet criteria for PPA and have mild behavioral changes, eye movement abnormalities or mild limb apraxia but who do not meet diagnostic criteria for, progressive supranuclear palsy or corticobasal syndrome respectively, will also be excluded.
* Subjects will be excluded from the study if they have any of the following genetic conditions which can increase the chance of cancer: Cowden disease, Lynch syndrome, hypogammaglobulinemia, Wiskott-Aldrich syndrome, and Down's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Josephs, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We leveraged data that had already been collected on healthy controls from our NIH funded Mayo Clinic Study of Aging (U01 AG006786). That study recruited healthy subjects of which 102 were controls, who had completed the identical tau-PET protocol with AV-1451 and MRI and clinical protocols. We selected a subset of 80 age and gender match healthy controls from the 102 for use in this study. These 80 participants were not consented or enrolled in this study.
Groups:
- Healthy Controls: Subjects from our NIH funded Mayo Clinic Study of Aging (U01 AG006786) who have completed the identical tau-PET protocol with AV-1451 and MRI and clinical protocols. These participants were not consented or enrolled in this study.
Period: Overall Study
Arm/Group | Tau PET Scan, F-18 AV 1451 | Healthy Controls
Started | 81 | 80
Completed | 75 | 80
Not Completed | 6 | 0
Not completed — Ineligible | 6 | 0

BASELINE CHARACTERISTICS:
Population: We leveraged data that had already been collected on healthy controls from our NIH funded Mayo Clinic Study of Aging (U01 AG006786). That study recruited healthy subjects of which 102 were controls, who had completed the identical tau-PET protocol with AV-1451 and MRI and clinical protocols. We selected a subset of 80 age and gender match healthy controls from the 102 for use in this study. These 80 participants were not consented or enrolled in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tau PET Scan, F-18 AV 1451 | Healthy Controls | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 46 | 43 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 95
  Male | 36 | 30 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 77 | 80 | 157
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 77 | 80 | 157
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 80 | 161

OUTCOME MEASURES:

1. Primary Outcome: Proportion of PPA Subjects That Showed Elevated Tau PET Binding Compared to Normal Controls
Description: The percentage of subjects who showed elevated tau PET binding in the following five categories: PPA Clinical Variant-logopenic (lvPPA), PPA Clinical Variant-semantic (svPPA), PPA Clinical Variant-agrammatic (agPPA), no clinical variant-healthy, and Unclassified Variant (PPA-U).
Time Frame: 1 week
Population: Subjects were subclassified into 1 of 5 categories based on clinical features. Classification for Tau PET Scan, F-18 AV 1451 arm: 4 lvPPA; 32 svPPA; 24 agPPA; 0 healthy; 9 PPA-U. Classification for Health Controls: 0 lvPPA; 0 svPPA; 0 agPPA; 80 healthy; 0 PPA-U.
Measure: Count of Participants; unit: Participants
Arm/Group | Tau PET Scan, F-18 AV 1451 | Healthy Controls
Number analyzed (Participants) | 69 | 80
Participants
  PPA Clinical Varient-logopenic (lvPPA): number analyzed (Participants) | 4 | 0
  PPA Clinical Varient-logopenic (lvPPA) | 3 | 0
  PPA Clinical Variant-semantic (svPPA): number analyzed (Participants) | 32 | 0
  PPA Clinical Variant-semantic (svPPA) | 17 | 0
  PPA Clinical Variant-agrammatic (agPPA): number analyzed (Participants) | 24 | 0
  PPA Clinical Variant-agrammatic (agPPA) | 5 | 0
  No Clinical Variant-healthy: number analyzed (Participants) | 0 | 80
  No Clinical Variant-healthy | 0 | 6
  PPA Clinical Variant-Unclassified (PPA-U): number analyzed (Participants) | 9 | 0
  PPA Clinical Variant-Unclassified (PPA-U) | 1 | 0

2. Secondary Outcome: Signature Patterns of Regional Tau PET Binding in Clinical PPA Variants
Description: To determine whether each of the three clinical PPA variants (logopenic (lvPPA), semantic (svPPA) and agrammatic (agPPA)) has a signature pattern of regional tau PET binding by measuring the level of tau PET binding in each PPA variant. 0=represents no specific uptake pattern; 1=specific uptake pattern
Time Frame: 1 Week
Population: 40 subjects were included in the analysis as there was enough data from these 40 subjects to address aim 2. Subjects were subclassified into 1 of 3 PPA variants based on clinical features. Classification: 14 lvPPA; 13 svPPA; 13 agPPA. Signature patterns of regional tau PET binding in clinical PPA variants were not measured in the Mayo Clinic Study of Aging trial, therefore the healthy controls arm does not apply to this outcome as no data exists for that arm.
Measure: Number; unit: units on a scale
Groups:
- Tau PET Scan, F-18 AV 1451: All subjects will received a Tau PET scan.
  F-18 AV 1451: Tau binding agent
Arm/Group | Tau PET Scan, F-18 AV 1451 | Healthy Controls
Number analyzed (Participants) | 40 | 0
units on a scale
  logopenic (lvPPA): number analyzed (Participants) | 14 | 0
  logopenic (lvPPA) | 1 |
  semantic (svPPA): number analyzed (Participants) | 13 | 0
  semantic (svPPA) | 1 |
  agrammatic (agPPA): number analyzed (Participants) | 13 | 0
  agrammatic (agPPA) | 1 |

3. Other Pre Specified Outcome: Variability in Patterns of Tau PET Binding
Description: To identify variability in patterns of tau PET binding using principal component (PC) analysis based on regional [18F]AV-1451 uptake to identify patterns between the three clinical variants: lvPPA, svPPA and agPPA independent of clinical diagnosis among PPA subjects. Two PCs were utilized to determine the number of participants who fell into the following 4 categories based on regional [18F]AV-1451 uptake patterns: low PC1/high PC2, low PC1/low PC2, high PC1/high PC2 and high PC1/low PC2. The first principal component (PC1) is a weighted sum of regional data where the weights are chosen so that PC1 has maximum variation across subjects. PC1 can be thought of as the "best" single-number summary of the regional data in a given modality. The second principal component (PC2) is a weighted sum of regional data with weight chosen so that (1) PC2 is completely uncorrelated with PC1 and (2) PC2 has maximum variation after accounting for PC1.
Time Frame: 1 Week
Population: 40 subjects were included in the analysis as there was enough data from these 40 subjects to address aim 3. Subjects were classified into groups based on uptake patterns. Classification: 5 Low PC1/High PC2; 10 Low PC1/Low PC2; 13 High PC1/High PC2, 12 High PC1/Low PC2.Variability in patterns of tau PET binding was not measured in the Mayo Clinic Study of Aging trial; therefore, the healthy controls arm does not apply to this outcome as no data exists for that arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tau PET Scan, F-18 AV 1451 | Healthy Controls
Number analyzed (Participants) | 40 | 0
Participants
  Low PC1/High PC2: number analyzed (Participants) | 5 | 0
  Low PC1/High PC2: lvPPA | 5 |
  Low PC1/High PC2: agPPA | 0 |
  Low PC1/High PC2: svPPA | 0 |
  Low PC1/Low PC2: number analyzed (Participants) | 10 | 0
  Low PC1/Low PC2: lvPPA | 9 |
  Low PC1/Low PC2: agPPA | 1 |
  Low PC1/Low PC2: svPPA | 0 |
  High PC1/High PC2: number analyzed (Participants) | 13 | 0
  High PC1/High PC2: lvPPA | 0 |
  High PC1/High PC2: agPPA | 0 |
  High PC1/High PC2: svPPA | 13 |
  High PC1/Low PC2: number analyzed (Participants) | 12 | 0
  High PC1/Low PC2: lvPPA | 0 |
  High PC1/Low PC2: agPPA | 12 |
  High PC1/Low PC2: svPPA | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 1 week.
Description: The participants in the healthy control arm did not receive the intervention and were not enrolled in the study. Adverse events were not collected on the healthy controls.
Arm/Group | Tau PET Scan, F-18 AV 1451 | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/0
Other Adverse Events (participants affected / at risk) | 0/81 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-10-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT02736695/Prot_000.pdf